CLINICAL TRIAL: NCT03307083
Title: Operating Check List During Consultation for Dental Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLIMAX
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Dental Implant
MeSH Terms: interventions — Foundations; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Check list FOR (Foundation for Oral Rehabilitation) — the surgeon uses this check list during the pre surgery consultation

SUMMARY:
Various studies showed how extent elements not directly linked to the state of the patient were involved in the failures in particular in surgery. That's why it's common to use check list system to avoid human mistakes or any other situation which could impact on the surgery.

Here the study 's aim is to assess a tool set up by the Foundation for Oral Rehabilitation ; it's a check list which cover all the treatment phases concerning dental implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient with dental implant surgery

Exclusion Criteria:

* refusing the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
number of adverst events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France